CLINICAL TRIAL: NCT07036484
Title: Supporting Couples' Perinatal Sexual Well-being: A Pilot Feasibility Study of the Introductory Modules of a Novel Prevention Program (STORK)
Brief Title: Supporting Couples' Perinatal Sexual Well-being: Testing the Introductory Modules of a Novel Prevention Program (STORK)
Status: Completed | Type: Observational
Sponsor: Dalhousie University (Other)
Collaborators: University of British Columbia (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-6719; 435-2023-0235 (Other Grant/Funding Number: Canadian Social Sciences and Humanities Research Council)
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2024-10

CONDITIONS: Pregnancy
Keywords: pregnancy; postpartum; perinatal; transition to parenthood; psychoeducation; internet intervention; prevention; sexual wellbeing; sexual health; couple

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Online program — We tested the feasibility of the introductory modules of an online couple-based program (STORK), designed to be grounded in empirically established risk and protective factors associated with couples' perinatal sexual well-being. STORK is a web-based program including psychoeducation and behavioral tasks to be completed by couples

SUMMARY:
Most new parents will experience changes to their sexual relationship during the perinatal period, yet no accessible prevention programs exist to support couples in navigating these changes. The goal of this observational study is to test the feasibility of the introductory modules of an online program (STORK) designed to promote perinatal sexual well-being in a sample of expectant couples. The main question it aims to answer is:

Is STORK a feasible and acceptable resource to support couples' perinatal sexual well-being? Couple participants who complete the first two modules of the STORK program will answer online survey questions and an interview about their experience with the program.

ELIGIBILITY:
Inclusion Criteria:

* both partners are at least 18 years of age
* both partners speak and read English fluently
* both partners live together and are in a relationship with each other for at least 1 year
* one partner is 12-25 weeks pregnant with both partner's first child

Exclusion Criteria:

- couples were instructed by a healthcare professional to avoid sexual activity during pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult couples who are in a cohabiting committed relationship with each other and are expecting their first baby (between 12-25 weeks gestation).
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2023-08-11 (Actual); Primary Completion 2023-12-08 (Actual); Study Completion 2023-12-08 (Actual)

PRIMARY OUTCOMES:
Acceptability | At entry (around 20 weeks gestation)
  After completing the initial STORK program's modules, couples self-reported on acceptability of the platform using 11 researcher-derived items modeled after prior similar work. Items assessed aspects such as enjoyment, overall organization, and amount of information for Module 0 and Module 1 using 7-point Likert-type response scales. Participants also provided open-ended suggestions for improvement.
Content and layout | At entry (around 20 weeks gestation)
  Participants self-reported on 9 researcher-derived items assessing the content and layout of information presented in the STORK program such as platform layout, clarity and appropriateness of content using 7-point Likert-type response scales. Three open-ended questions asked about areas that were covered well, areas of improvement, and confusing terms/ideas.
Functionality | At entry (around 20 weeks gestation)
  Two researcher-derived items assessed ease of navigation and the relevance of graphics (i.e., images/videos) using 7-point Likert-type response scales; an open-ended question asked about specific suggestions to functionality of the platform.
Inclusivity | At entry (around 20 weeks gestation)
  Participants self-reported on their perceptions regarding inclusivity of the platform using 4 researcher-derived items completed on a 7-point Likert-type response scales. One open-ended question asked about specific suggestions to improve inclusivity of the program.
Time commitment | At entry (around 20 weeks gestation)
  Participants self-reported how long it took them to complete the modules, and whether they considered this amount of time reasonable using a dichotomic (yes/no) item; if they responded negatively, then they were invited to provide reasons using an open-ended question.
Feasibility of the program's introductory modules - semi structured interview | At entry (around 20 weeks gestation)
  After completing the module, a semi-structured interview was conducted. The interview included open-ended questions about the web platform, as well as specific questions regarding its content, relevancy, clarity, organization, aesthetics, navigation, and functionality.

CONTACTS AND LOCATIONS:
Overall Officials: Natalie O Rosen, Ph.D., Principal Investigator — Dalhousie University, Canada; Samantha J Dawson, Ph.D., Principal Investigator — University of British Columbia, Canada; Inês M Tavares, Ph.D., Principal Investigator — Lusófona University, Portugal
Locations (1):
- Dalhousie University, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No